CLINICAL TRIAL: NCT04525703
Title: Intervention Feasibility Study - Fatherhood After Prison: Healthy Children and Families
Brief Title: Pathways for Parents After Incarceration Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0144; A488200 (Other: UW Madison); L&S/SOCIAL WORK/SOC WORK (Other: UW Madison); 4R00HD081273-03 (NIH); Protocol Version 7/8/2021 (Other: HSIRB, UW Madison)
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Parenting; Development, Child; Behavior
Keywords: incarceration; antisocial behavior; family; child development
MeSH Terms: conditions — Behavior; Antisocial Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pathways for Parents (Experimental)
  Interventions: Behavioral: Pathways for Parents after Incarceration

INTERVENTIONS:
Behavioral: Pathways for Parents after Incarceration — The Pathways for Parents after Incarceration program uses eight key lessons, including topics on effective listening, speaking, and problem-solving skills, lessons on emotion regulation, and issues surrounding family engagement. The program (both classroom and therapeutic peer support) will be offered virtually and weekly for 8 continuous weeks.

SUMMARY:
The purpose of this study is to learn how to better support fathers and their families after incarceration. It will test an intervention that promotes healthy development for children of previously incarcerated fathers and the caregivers of their children for empirical promise through a pilot feasibility trial. The aims of the pilot are to demonstrate: a) client acceptance of the treatment (e.g., retention), b) ability to recruit sufficient numbers of participants, and c) feasibility of delivery with the clients and therapists in the designated treatment settings. About 15 families (15 fathers, 15 caregivers, and 15-20 children, totaling 45-50 participants) will be in the study.

DETAILED DESCRIPTION:
The purpose of the overall study, Promoting Healthy Development among Children of Fathers with Antisocial Behavior, is to build and test a preventive family-focused intervention in a feasibility study that promotes healthy development for children of previously incarcerated fathers and the caregivers of their children. The study has three specific aims, two of which have already been completed. The first was to conduct secondary data analyses to explore a series of questions that explored topics including fathers' history of antisocial behavior and criminality, children's psycho-social and behavioral health outcomes, father engagement and parenting behavior, maternal parenting practices, quality of parental relationship, and extended family involvement. The second aim included conducting semi-structured interviews with fathers, mothers, and relatives to improve understanding of the barriers to father engagement and challenges that families face as fathers return to the community following incarceration.

To that end, this protocol situates itself within the third and final aim, that of specifying treatment procedures (e.g., develop manuals, select measures, specify therapist training and adherence procedures) and establishing feasibility of the intervention (e.g., recruitment, enrollment, fidelity, adherence, retention, and safety). Specifically, this protocol is in regard to the feasibility of the intervention. The purpose is to test the intervention for empirical promise through a pilot feasibility trial. The aims of the pilot are to demonstrate: a) client acceptance of the treatment (e.g., retention), b) ability to recruit sufficient numbers of participants, and c) feasibility of delivery with the clients and therapists in the designated treatment settings.

The family intervention is based in a family systems model that includes all members of the family. Multiple family groups are used because previous research has found they are efficient forms of service delivery, build social support among participants, and improve parent-child interactions. Feasibility of the pilot must include all participants anticipated in the program model to test strategies, logistics, and measures. Drawing from the framework of dissemination and implementation science, another central purpose of the pilot is to refine the operational methods that will facilitate translation and implementation in the future should the intervention be found efficacious and effective. This pilot will answer questions that are pertinent to intervention development, as well as the success of dissemination and implementation in the future.

The Intervention:

Pathways for Parents after Incarceration (P4P) is a community-based program that seeks to equip fathers with the skills both for positive father engagement and reentry success. It uses a manualized curriculum that is adapted from a prison-based program, Parenting Inside Out (PIO). PIO is an evidence-based, cognitive-behavioral parent management skills training program created for incarcerated parents through a six-year collaboration of scientists, policy makers, practitioners, and instructional designers. Both the information in the program and the way that information is presented were informed by knowledge derived from research and practice. Extracted from the full 90-hour version, the Pathways for Parents after Incarceration program uses eight key lessons from the original version that have been identified by the research team and those with lived experience as being most beneficial to them. These include topics on effective listening, speaking, and problem-solving skills, lessons on emotion regulation, and issues surrounding family engagement. The course is led by 2 parent coaches who will be interviewed by program leaders and formally trained to deliver PIO by the PIO parent organization, The Pathfinder Network. The classroom-based PIO sessions will be delivered over 8 weeks in two-hour sessions.

In addition to the classroom component that PIO provides, the program will offer a therapeutic component. Weekly, those receiving services from Pathways for Parents after Incarceration will be invited to take part in a peer support group-style group session led by an esteemed provider within the community, Anesis Family Therapy. This component of the program is rooted in systems therapy and uses narrative therapy, trauma focused cognitive therapy, and motivational interviewing techniques. This aspect promotes fathers' and caregivers' ability to identify their values and skills so they can effectively confront the challenges (both instrumental and relational) that they face during their reentry period and as family members working to support the fathers. These sessions run for 45 minutes following the classroom portion.

The program (both classroom and therapeutic peer support) will be offered weekly on a weekday evening for 8 continuous weeks (the 9th week will be a class graduation/celebration). The sessions will be offered virtually to accommodate safety protocols related to the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria (fathers):

* being able to speak and read English
* having at least one child between the ages of 3 and 17-years-old
* having been released from incarceration within the last 5 years (from county jail or state/federal prison)
* play a parenting role in at least some way (e.g., residence, contact, phone, etc.)

Inclusion Criteria (caregivers):

* able to speak and read English
* at least 18-years-old

Exclusion Criteria:

* have been convicted of a crime against any of his children
* are prevented from having contact with their child

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pajarita Charles, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Pathways for Parents after Incarceration Program study was conducted between September 2020 and March 2022 during the COVID-19 pandemic.
Pre-assignment Details: 51 Fathers were assessed for eligibility, 43 were eligible, 21 consented and started the study.
Groups:
- Caregivers; Fathers; Children: Pathways for Parents after Incarceration: The Pathways for Parents after Incarceration program uses eight key lessons, including topics on effective listening, speaking, and problem-solving skills, lessons on emotion regulation, and issues surrounding family engagement. The program (both classroom and therapeutic peer support) will be offered virtually and weekly for 8 continuous weeks.
Period: Overall Study
Arm/Group | Caregivers | Fathers | Children
Started | 12 | 21 | 15
Completed Baseline Interview | 12 | 21 | 15
Attended Any of the P4P Program | 9 | 16 | 11
Completed P4P Program | 7 | 12 | 9
Completed Post Intervention Survey | 7 | 12 | 9
Completed 3-month Follow up Survey | 6 | 6 | 7
Completed | 6 | 6 | 7
Not Completed | 6 | 15 | 8
Not completed — Lost to Follow-up | 6 | 15 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caregivers | Fathers | Children | Total
Number analyzed (Participants) | 12 | 21 | 15 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 15 | 15
  Between 18 and 65 years | 11 | 21 | 0 | 32
  >=65 years | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 8 | 20
  Male | 0 | 21 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 4 | 10
  Not Hispanic or Latino | 9 | 18 | 11 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 12 | 6 | 24
  White | 3 | 6 | 4 | 13
  More than one race | 2 | 2 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 21 | 15 | 48
Time Since Incarceration [Mean (Standard Deviation); unit: months] | NA (NA) — Caregivers Not Incarcerated | 8 (13.94) | NA (NA) — Children Not Incarcerated | 8 (13.94)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Fathers and Caregivers Who Consent
Description: The feasibility of this approach will in part be measured by successful recruitment of participants from this population. This is measured by the proportion of eligible fathers and caregivers who consent to study participation and enrollment.
Time Frame: baseline
Population: 43 Fathers were eligible, 23 consented and started the study
Measure: Number; unit: proportion of participants
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 43 | 12
proportion of participants | 0.49 | 1.0

2. Primary Outcome: Proportion of Enrolled Fathers and Caregivers Who Complete Entire Intervention
Description: The feasibility of this approach will in part be measured by the retention of participants in this intervention. This is measured by the proportion of enrolled fathers and caregivers who participate in the first intervention class (after baseline) and complete entire intervention.
Time Frame: up to 9 weeks
Population: This combined criteria (enrolled AND participated in the first intervention class) changes the baseline N to something smaller (n=16, not n=21)
Measure: Number; unit: proportion of participants
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 16 | 12
proportion of participants | 0.75 | 0.58

3. Primary Outcome: Provider Adherence Measured by the Parenting Inside Out Group Observation Feedback Form Score
Description: Adherence is measured using the Parenting Inside Out (PIO) Group Observation Feedback Form to assess program integrity and fidelity to the model. This is a 35-item survey that assesses 5 domains: curriculum delivery and fidelity; facilitation skills, behavior support and group management; interpersonal skills, and PIO specific items. Each item is scored on a scale of 1-5 where 1 is remediation needed, 2 is growth area, 3 is developing, 4 is effective, and 5 is highly effective. Average scores from each domain are reported for a total possible range of scores 1-5, higher scores indicate better adherence.
Time Frame: up to 9 weeks
Population: Team stopped collecting this survey after 3 responses as it was determined to be burdensome for the participant and not useful for the investigation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pathways for Parents
Number analyzed (Participants) | 3
score on a scale
  Overall Fidelity | 4.46 (0.16)
  Curriculum Delivery & Fidelity Subscale | 4.57 (0.14)
  Facilitation Skills Subscale | 4.55 (0.04)
  Behavior Support and Group Management Subscale | 4.86 (0.14)
  Interpersonal Skills Subscale | 5.00 (0.00)
  PIO Specific Skills Subscale | 4.17 (0.32)

4. Primary Outcome: Acceptability of Intervention Assessed by Providers
Description: Acceptability is assessed by interventionists using an overall rating of the content delivered to participants each week.
  The overall score is rated on a scale of 1=poor to 10=excellent, with higher scores indicating greater acceptability.
Time Frame: up to 9 weeks
Population: Providers were not consented to the study, but were surveyed for acceptability of the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Providers: Providers for the Pathways for Parents after Incarceration Program.
Arm/Group | Providers
Number analyzed (Participants) | 2
score on a scale | 8.43 (0.37)

5. Primary Outcome: Self-Perceived Helpfulness of the Program for the Participant
Description: Acceptability and usefulness of the intervention is assessed in part by a series of questions that ascertain perceived helpfulness of program for the participant.
  How helpful was the parenting program for you? 1= Not at all helpful, 2=A little helpful, 3=Somewhat helpful, 4=Quite helpful, 5=Very helpful
Time Frame: up to 21 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale | 4.67 (0.65) | 4.71 (0.49)

6. Primary Outcome: Participant-Perceived Helpfulness of the Program for the Participant's Child
Description: Acceptability and usefulness of the intervention is assessed in part by a series of questions that ascertain perceived helpfulness of program for the participant.
  "Overall, do you think your participation in this program has had any effect on your child?" 1=has had a very negative effect, 5=has had a very positive effect.
Time Frame: up to 21 weeks
Population: There are missing data from 2 participants in the Fathers group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caregiver: Pathways for Parents after Incarceration: The Pathways for Parents after Incarceration program uses eight key lessons, including topics on effective listening, speaking, and problem-solving skills, lessons on emotion regulation, and issues surrounding family engagement. The program (both classroom and therapeutic peer support) will be offered virtually and weekly for 8 continuous weeks.
Arm/Group | Fathers | Caregiver
Number analyzed (Participants) | 10 | 7
score on a scale | 3.90 (0.57) | 4.43 (0.53)

7. Primary Outcome: Acceptability of Intervention Assessed by Participant Recommendation
Description: Acceptability and usefulness of the intervention is assessed in part by a series of questions that ascertain whether participants would recommend the program to other people.
  Would you recommend this program to other parents? 1=Strongly recommend, 2=Recommend, 3=Neutral, 4=Not recommend, 5=Strongly not recommend
Time Frame: up to 21 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale | 4.83 (0.39) | 5.00 (0.00)

8. Primary Outcome: Acceptability of Intervention Assessed by Parent Satisfaction
Description: Acceptability and usefulness is assessed by a series of questions that ascertain parent satisfaction.
  Q: How much has the Parenting Inside Out classes changed how happy and satisfied you are with being a parent to your child? 1=none, 2=A little, 3=Some, 4=A lot, 5=Very much
Time Frame: up to 21 weeks
Population: One participant in the Fathers group did not answer the survey item.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 11 | 7
score on a scale | 4.64 (0.67) | 4.57 (0.53)

9. Secondary Outcome: Inventory of Family Feelings Score
Description: Family interactions & relationships will be assessed with the 38-item Inventory of Family Feelings to assess fathers' and caregivers' perceptions of their relationship with another and with their children. Scores range from 0-38, with higher scores indicating more positive affect toward family members and lower scores reflecting conflicted relationships.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 16.0 (1.58) | 16.14 (2.06)
  Post-test | 14.17 (1.98) | 15.57 (0.57)

10. Secondary Outcome: Coparenting Relationship Scale Score: Undermining Subscale
Description: The Undermining subscale of the Coparenting Relationship Scale contains 3-items, scored on a scale of 1=strongly disagree to 5=strongly agree. Change in summed score will be reported (between 3-15) with lower scores indicative of a stronger coparenting relationship.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 6.6 (0.83) | 7.0 (0.88)
  Post-test | 6.8 (1.0) | 6.9 (1.4)

11. Secondary Outcome: Coparenting Relationship Scale Score: Alliance Subscale
Description: The Alliance subscale of the Coparenting Relationship Scale contains 5-items, scored on a scale of 1=strongly disagree to 5=strongly agree. Change in summed score will be reported (between 5-25) with higher scores indicative of a stronger coparenting relationship.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 18.7 (1.5) | 21.9 (1.5)
  Post-test | 18.8 (1.6) | 21.4 (1.3)

12. Secondary Outcome: Coparenting Relationship Scale Score: Gatekeeping Subscale
Description: The Gatekeeping subscale of the Coparenting Relationship Scale contains 3 items, scored on a scale of 1=strongly disagree to 5=strongly agree. Change in summed score will be reported (between 3-15) with lower scores are indicative of a stronger coparenting relationship.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 5.5 (0.61) | 5.3 (0.75)
  Post-test | 5.2 (0.83) | 3.7 (0.47)

13. Secondary Outcome: Kansas Parenting Satisfaction Scale Score
Description: Parenting Satisfaction will be assessed with a 3-item scale, Kansas Parenting Satisfaction Scale. Items are scored on a scale of 1=extremely dissatisfied to 7=extremely satisfied. Change in summed score will be reported (between 3-21) with higher scores indicative of higher levels of parenting satisfaction.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 16.8 (0.84) | 16.0 (1.45)
  Post-test | 15.1 (1.4) | 16.4 (1.31)

14. Secondary Outcome: Parenting Sense of Competence Scale Score
Description: Parenting competence assessed with the 17-item Parenting Sense of Competence Scale. Items are scored on a scale of 1=strongly disagree to 6=strongly agree. Scores range from 17-102, with higher scores indicative of a stronger sense of competence, satisfaction and efficacy.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 78.8 (2.1) | 74.7 (5.12)
  Post-test | 76.4 (2.1) | 76.7 (5.12)

15. Secondary Outcome: Alliance Measure Score
Description: Parenting alliance is assessed with the 20-items self-report Parenting Alliance Measure. Items are scored on a 5-point rating scale ranging from 1=strongly disagree to 5=strongly agree. Change in summed score will be reported (between 20-100), with higher scores reflecting stronger coparenting alliances between people.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 80.1 (4.8) | 87.1 (5.1)
  Post-test | 82.4 (5.1) | 83.4 (5.3)

16. Secondary Outcome: Child-Parent Relationship Scale (CPRS) Score: Conflict Subscale
Description: Assessed with the 15-item Child-Parent Relationship Scale-Short Form to assess perceptions of participants' relationship with their children. The Conflict subscale contains 8-items, scored on a scale of 1=definitely does not apply to 5=definitely applies. Change in summed scores (between 8 and 40) for each subscale over time will be reported, higher scores on each subscale (closeness, conflict) indicative of higher levels of each dimension.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 19.3 (1.7) | 17.86 (1.4)
  Post-test | 18.3 (1.7) | 16.1 (1.5)

17. Secondary Outcome: Child-Parent Relationship Scale (CPRS) Score: Closeness Subscale
Description: Assessed with the 15-item Child-Parent Relationship Scale-Short Form to assess perceptions of participants' relationship with their children. The Closeness subscale contains 7-items, scored on a scale of 1=definitely does not apply to 5=definitely applies. Change in summed scores (between 7 and 35) for each subscale over time will be reported, higher scores on each subscale (closeness, conflict) indicative of higher levels of each dimension.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 30.4 (1.3) | 31.1 (0.74)
  Post-test | 30.2 (1.4) | 29.43 (2.58)

18. Secondary Outcome: Cohen Perceived Stress Scale Score
Description: Stress will be assessed with the 10-item Cohen Perceived Stress Scale. Items are scored on a scale of 0=never to 4=very often. Change in summed score (between 0-40) will be reported, with higher scores reflecting higher levels of stress experienced by the participant.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 34.2 (2.5) | 33.57 (2.99)
  Post-test | 32.0 (1.8) | 33.71 (2.92)

19. Secondary Outcome: Center for Epidemiologic Studies Depression (CESD) Depression Scale Score
Description: Depression will be assessed with the CESD Depression Scale. Items are scored on a scale of 0=rarely or none of the time (or less than 1 day) to 3=most or all of the time (5-7 days). Change in summed score (between 0-60) will be reported, with higher scores indicating the presence of more depression symptomology.
Time Frame: Baseline (pre-test), 9 weeks (post-test)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Fathers | Caregivers
Number analyzed (Participants) | 12 | 7
score on a scale
  Pre-test | 15.0 (2.5) | 9.71 (2.9)
  Post-test | 12.8 (2.2) | 10.86 (3.81)

ADVERSE EVENTS:
Time Frame: up to 21 weeks
Arm/Group | Caregivers | Fathers | Children
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/21 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/21 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/21 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT04525703/Prot_SAP_001.pdf
  • Informed Consent Form (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT04525703/ICF_000.pdf